CLINICAL TRIAL: NCT02838615
Title: Comparison of Lumbar Epidural Steroid Injection: Transforaminal vs. Parasagittal Interlaminar Approach
Brief Title: Comparison of Transforaminal vs. Parasagittal Interlaminar Epidural Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Associate professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-05-029
Record Dates: First submitted 2016-05-25; First posted 2016-07-20 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Spinal Stenosis
Keywords: spinal stenosis; epidural steroid injection
MeSH Terms: conditions — Spinal Stenosis | interventions — Dexamethasone; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- epidural steroid injection (Active Comparator): TF epidural steroid (dexamethasone) injection
  Interventions: Procedure: epidural steroid (dexamethasone) injection
- IL epidural steroid injection (Active Comparator): PS interlaminar epidural steroid(dexamethasone) injection
  Interventions: Procedure: epidural steroid (dexamethasone) injection

INTERVENTIONS:
Procedure: epidural steroid (dexamethasone) injection — spinal injections performed in epidural space to relieve chronic low back pain or leg pain

SUMMARY:
The purpose of this study is to compare the clinical efficacy, incidence of ventral epidural spreading and provocation of concordant paresthesia, amount of radiation exposure and total procedure time between transforaminal and parasagittal interlaminar epidural injection.

DETAILED DESCRIPTION:
Participants were randomly allocated to receive either parasagittal interlaminar or transforaminal ESI.

Investigators obtained clinical data including age, gender, duration of symptoms, predominant symptoms (axial pain vs. leg pain), severity of neurogenic intermittent claudication (NIC) and degree of depression. Depression was assessed by the Korean version of the Beck Depression Inventory (BDI). The BDI is a standardized questionnaire to assess cognitive, affective, and somatic symptoms of depression. All data were obtained before performing ESI.Data about anterior epidural spreading and presence of concordant pain provocation were obtained during fluoroscopic guided parasagittal interlaminar or transforaminal ESI. Also total procedure time and amount of radiation exposure were checked. Investigators observed the epidural spread pattern after a 2 ml injection of contrast material, confirmed anterior epidural spread with a lateral view, and asked the participants if they had any concordant pain provocation or not. The participants were asked if the pain was in the same distribution as their original pain (concordant) or dissimilar or absent in both quality and location.

Investigators used the numerical rating scale (NRS) as well as the Korean version of the Oswestry Disability Index (ODI) to evaluate clinical efficacy in terms of reducing pain and functional improvement at pretreatment and 2 weeks after the ESI series. ESI was performed twice with a 2 weeks interval before the final treatment outcome evaluation with the NRS and ODI. All patients reported average severity of their symptoms over the previous 1 week. A score of 0 on the NRS represents no pain, and a score of 10 represents the worst pain imaginable. The Korean version of the ODI (0-50) was used to assess functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* central spinal stenosis
* herniated nucleus pulposus.

Exclusion Criteria:

* Lateral spinal stenosis
* Internal disc disruption

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy | 2 weeks after study completion
  Numerical rating scale

SECONDARY OUTCOMES:
Intervention related time | 1 minutes after the completion of the intervention
  time required to complete the intervention
Exposed radiation amount during intervention | 1 minutes after the completion of the intervention
  Exposed radiation amount during intervention

IPD SHARING:
Plan to Share IPD: No